CLINICAL TRIAL: NCT02262260
Title: A Randomized, Open-label Non-inferiority Study to Compare Safety and Efficacy of Labeled Versus Wait and Extend Regimen of Lucentis (Ranibizumab) in Turkish Patients With Visual Impairment Due to Diabetic Macular Edema.
Brief Title: Compare Safety/Efficacy of Labeled vs Wait-Extend Regimen of Lucentis in Turkish Patients With VI Due to DME
Acronym: SALUTE-D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002DTR01
Record Dates: First submitted 2014-08-27; First posted 2014-10-13 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-03

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic macular edema, DME, ranibizumab, wait and extend
MeSH Terms: interventions — DMAC2L protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab labeled regime arm (Experimental): Ranibizumab (Anti VEGF) 0.5mg treatment will be given monthly and will be continued until maximum visual acuity is achieved (the patient's visual acuity is stable for three consecutive monthly assessments performed while on ranibizumab treatment). Thereafter patients should be monitored monthly for visual acuity. Treatment will be resumed when monitoring indicates loss of visual acuity due to DME. Monthly injections should then be administered until stable visual acuity is reached again for three consecutive monthly assessments (implying a minimum of two injections). The interval between two doses should not be shorter than 1 month
  Interventions: Drug: Labeled regime arm
- Ranibizumab wait and Extend regime arm (Experimental): Ranibizumab (Anti VEGF) 0.5 mg will be injected subsequently at baseline, month 1 and 2. After the three initial loading doses, patients will be called for the control visits 1 month later. If the visual acuity has reached a stable level and there is no sign of edema on OCT, patients will not receive intravitreal injection and will be called to come back 6 weeks later. The interval is increased by 2 weeks until a maximum of 8 weeks as long as the patient presents as stable regarding visual acuity, central retinal thickness and clinical findings. If there is a negative change, the interval is shortened back to 4 weeks.
  Interventions: Drug: Wait and Extend regime arm

INTERVENTIONS:
Drug: Labeled regime arm — Treatment will be given monthly and will be continued until maximum visual acuity is achieved (the patient's visual acuity is stable for three consecutive monthly assessments performed while on ranibizumab treatment). Thereafter patients should be monitored monthly for visual acuity. Treatment will be resumed when monitoring indicates loss of visual acuity due to DME. Monthly injections should then be administered until stable visual acuity is reached again for three consecutive monthly assessments (implying a minimum of two injections). The interval between two doses should not be shorter than 1 month.
  Other Names: Arm 1
  Arms: Ranibizumab labeled regime arm
Drug: Wait and Extend regime arm — Lucentis (ranibizumab) 0.5 mg will be injected subsequently at baseline, month 1 and 2. After the three initial loading doses, patients will be called for the control visits 1 month later. If the visual acuity has reached a stable level and there is no sign of edema on OCT, patients will not receive intravitreal injection and will be called to come back 6 weeks later. The interval is increased by 2 weeks until a maximum of 8 weeks as long as the patient presents as stable regarding visual acuity, central retinal thickness and clinical findings. If there is a negative change, the interval is shortened back to 4 weeks.
  Other Names: Arm 2
  Arms: Ranibizumab wait and Extend regime arm

SUMMARY:
To explore a more clinical feasible treatment regime with ranibizumab for DME to provide satisfactory treatment effect with a lower number of visits and injections.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is the most common endocrine disease in developed countries, with prevalence estimates ranging between 2 to 5% of the world's population. Diabetic retinopathy (DR) and diabetic macular edema (DME) are common microvascular complications in patients with diabetes and may have a sudden and debilitating impact on visual acuity (VA), eventually leading to blindness. DME is a frequent manifestation of DR and is the major cause of visual loss in patients with DR. If left untreated, >50% of patients lose >2 lines of visual acuity (VA) within 2 years. DME mostly affects the working-age population, imposing a significant burden both on society and on individual patients - a burden that is expected to increase with the rising prevalence of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* M or F patients >18 years of age who have signed an informed consent
* Patients with Type 1 or Type 2 DM (according to ADA or WHO guidelines) with HbA1c not more than 12.0% at screening (Visit 1). Patients should be on diet, exercise, and/or pharmacological treatment for diabetes.
* Patients with visual impairment due to focal or diffuse macular edema with center involvement in at least one eye, as demonstrated with color fundus photography, fluorescein angiography and OCT within 28 days of the baseline treatment. If both eyes are eligible, the one with the worse visual acuity, as assessed at Visit 1, will be selected for study treatment unless, based on medical reasons, the investigator deems the other eye the more appropriate candidate for study treatment. The study eye must fulfill the following criteria at Visit 1:
* BCVA score between 78 and 39 letters, inclusively, using ETDRS-like visual acuity testing charts at a testing distance of 4 meters (approximate Snellen equivalent of 20/32 to 20/160)
* Decrease in vision is due to DME and not due to other causes, in the opinion of the investigator

Exclusion Criteria

* Concomitant conditions in the study eye according to defined criteria such as infection, inflammation, uncontrolled glaucoma
* Active PDR in the study eye or evidence of vitreomacular traction in either eye
* Patients who are monocular or have a BCVA score in the non-study eye (fellow eye) £ 24 letters at Visit 1
* Concomitant systemic condition according to defined criteria, eg. history of stroke, uncontrolled diabetes, renal failure, unsatisfactory controlled hypertension
* Use of other investigational drugs within 5 half-lives of enrollment, or within 30 days until the expected PD effect has returned to baseline, whichever is longer.
* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of study treatment.

Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-12-12 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Labeled Regime Arm | Wait and Extend Regime Arm
Started | 45 | 42
Completed | 34 | 32
Not Completed | 11 | 10
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal of consent | 4 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol deviation | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Labeled Regime Arm | Wait and Extend Regime Arm | Total
Number analyzed (Participants) | 45 | 42 | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61 (9.93) | 59.5 (9.68) | 60.3 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 29 | 27 | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in "Best-corrected Visual Acuity" at Month 12
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (ETDRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of ETDRS is 0 to 100 letters. A positive average change from baseline of BCVA indicates improvement
Time Frame: 12 months
Population: Study completers- The patients who have completed 12 months of treatment and follow-up are defined as Study Completers.
Measure: Mean (Standard Error); unit: Letters
Arm/Group | Labeled Regime Arm | Wait and Extend Regime Arm
Number analyzed (Participants) | 34 | 32
Letters | 76.44 (1.78) | 73.09 (1.68)
Statistical Analysis 1: Comparison: Labeled Regime Arm vs Wait and Extend Regime Arm; Test type: Non-Inferiority — In order to demonstrate that the "wait and extend" regimen of ranibizumab is non-inferior to the posology described in the prescribing information, mean change in BCVA at month 12 from the baseline visit were determined for both treatment groups, and a comparison was made between the two groups using the Independent Samples t-test; p = 0.5, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Mean Change in Central Retinal Thickness (CRT)
Description: CRT was assessed by Optical Coherence Tomography (OCT).
Time Frame: 12 months
Population: Study completers- The patients who have completed 12 months of treatment and follow-up are defined as Study Completers.
Measure: Mean (Standard Error); unit: Micrometers
Arm/Group | Labeled Regime Arm | Wait and Extend Regime Arm
Number analyzed (Participants) | 34 | 32
Micrometers | 315.7 (15.07) | 348.9 (16.54)
Statistical Analysis 1: Comparison: Labeled Regime Arm vs Wait and Extend Regime Arm; Test type: Non-Inferiority — In order to demonstrate that the "wait and extend" regimen of ranibizumab is non-inferior to the posology described in the prescribing information, mean change in Central Retinal Thickness determined with Optical Coherence Tomography for both eyes were calculated for both groups and were compared using the Mann Whitney u test; p = 0.082, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Mean Number of Injections
Description: Mean number of injections over a 12-month treatment period
Time Frame: 12 months
Population: Study completers- The patients who have completed 12 months of treatment and follow-up are defined as Study Completers. Statistical analysis not performed for the injection numbers
Measure: Mean (Standard Error); unit: Injections
Arm/Group | Labeled Regime Arm | Wait and Extend Regime Arm
Number analyzed (Participants) | 34 | 32
Injections | 7.4 (0.44) | 7.5 (0.44)

4. Secondary Outcome: Mean Number of Visits
Description: Mean number of visits over a 12-month treatment period
Time Frame: 12 months
Population: Study completers- The patients who have completed 12 months of treatment and follow-up are defined as Study Completers. Statistical analysis not performed to compare visits
Measure: Mean (Standard Error); unit: Number of visits
Arm/Group | Labeled Regime Arm | Wait and Extend Regime Arm
Number analyzed (Participants) | 34 | 32
Number of visits | 11.2 (0.19) | 10.2 (0.24)

5. Secondary Outcome: Proportion of Patients Who Gained ≥5 Letters
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An increased score indicates improvement in acuity. This outcome assessed the number of participants who had improvement of ≥5 letters of visual acuity at month 12 as compared with baseline
Time Frame: 12 months
Population: Study completers- The patients who have completed 12 months of treatment and follow-up are defined as Study Completers
Measure: Number; unit: Participants
Arm/Group | Labeled Regime Arm | Wait and Extend Regime Arm
Number analyzed (Participants) | 34 | 32
Participants | 29 | 22
Statistical Analysis 1: Comparison: Labeled Regime Arm vs Wait and Extend Regime Arm; Test type: Non-Inferiority — Comparison was made between the two groups using the Independent Samples t-test; p = 0.095, Chi-squared

6. Secondary Outcome: Proportion of Patients Who Gained ≥10 Letters
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An increased score indicates improvement in acuity. This outcome assessed the number of participants who had improvement of ≥10 letters of visual acuity at month 12 as compared with baseline
Time Frame: 12 months
Population: Study completers- The patients who have completed 12 months of treatment and follow-up are defined as Study Completers
Measure: Number; unit: Participants
Arm/Group | Labeled Regime Arm | Wait and Extend Regime Arm
Number analyzed (Participants) | 34 | 32
Participants | 23 | 15
Statistical Analysis 1: Comparison: Labeled Regime Arm vs Wait and Extend Regime Arm; Test type: Non-Inferiority — comparison was made between the two groups using the Independent Samples t-test; p = 0.072, Chi-squared

7. Secondary Outcome: Proportion of Patients Who Gained ≥15 Letters
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An increased score indicates improvement in acuity. This outcome assessed the number of participants who had improvement of ≥15 letters of visual acuity at month 12 as compared with baseline
Time Frame: 12 months
Population: Study completers- The patients who have completed 12 months of treatment and follow-up are defined as Study Completers
Measure: Number; unit: Participants
Arm/Group | Labeled Regime Arm | Wait and Extend Regime Arm
Number analyzed (Participants) | 34 | 32
Participants | 12 | 10
Statistical Analysis 1: Comparison: Labeled Regime Arm vs Wait and Extend Regime Arm; Test type: Non-Inferiority — comparison was made between the two groups using the Independent Samples t-test; p = 0.466, Chi-squared

ADVERSE EVENTS:
Time Frame: 12 month study
Groups:
- Labeled Treatment Arm: Treatment will be given monthly and will be continued until maximum visual acuity is achieved (the patient's visual acuity is stable for three consecutive monthly assessments performed while on ranibizumab treatment). Thereafter patients should be monitored monthly for visual acuity. Treatment will be resumed when monitoring indicates loss of visual acuity due to DME. Monthly injections should then be administered until stable visual acuity is reached again for three consecutive monthly assessments (implying a minimum of two injections). The interval between two doses should not be shorter than 1 month
- Wait and Extend Regimen Arm: Lucentis (ranibizumab) 0.5 mg will be injected subsequently at baseline, month 1 and 2. After the three initial loading doses, patients will be called for the control visits 1 month later. If the visual acuity has reached a stable level and there is no sign of edema on OCT, patients will not receive intravitreal injection and will be called to come back 6 weeks later. The interval is increased by 2 weeks until a maximum of 8 weeks as long as the patient presents as stable regarding visual acuity, central retinal thickness and clinical findings. If there is a negative change, the interval is shortened back to 4 weeks.
Arm/Group | Labeled Treatment Arm | Wait and Extend Regimen Arm
All-Cause Mortality (participants affected / at risk) | 1/45 | 0/42
Serious Adverse Events (participants affected / at risk) | 10/45 | 7/42
Other Adverse Events (participants affected / at risk) | 12/45 | 9/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Labeled Treatment Arm (N=45) | Wait and Extend Regimen Arm (N=42)
Angina pectoris (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1
Vitreous hemorrhage (Eye disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Labeled Treatment Arm (N=45) | Wait and Extend Regimen Arm (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 1 | 1
Itchy eyes (Eye disorders) | 1 | 0
Ocular hyperemia (Eye disorders) | 2 | 1
Vitreoretinal traction syndrome (Eye disorders) | 1 | 1
Vitreous hemorrhage (Eye disorders) | 0 | 1
Vitreous opacity (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2
Gastric spasm (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Ocular hyperemia (Gastrointestinal disorders) | 1 | 0
Gall bladder stone (Hepatobiliary disorders) | 0 | 1
Gallbladder inflammation (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Adenovirus infection (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 0 | 1
Foot infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Increased intraocular pressure (Investigations) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Gallbladder papillary adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tinnitus (Nervous system disorders) | 1 | 0
Impaired renal function (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT02262260/SAP_000.pdf
  • Study Protocol (2016-04-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT02262260/Prot_001.pdf